CLINICAL TRIAL: NCT05973786
Title: A Randomised, Controlled Trial to Investigate the Effect of a Six Week Intensified Pharmacological Treatment for Bipolar Depression Compared to Treatment as Usual in Subjects Who Had a First-time Treatment Failure on Their First-line Treatment.
Brief Title: The Effect of a Six Week Intensified Pharmacological Treatment for Bipolar Depression Compared to Treatment as Usual in Subjects Who Had a First-time Treatment Failure on Their First-line Treatment.
Acronym: INTENSIFY BD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Inge Winter (Other)
Collaborators: Universität Münster (Other)
Responsible Party: Sponsor-Investigator, Dr. Inge Winter, Principal Investigator, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-506605-19-00 (EU CT#)
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Escitalopram; Sertraline; Venlafaxine Hydrochloride; Lithium; Quetiapine Fumarate; Bupropion

STUDY DESIGN:
Intervention Model Description: Parallel randomization to the 2 arms, treatment as usual (TAU) or early-intensified pharmacological treatment (EIPT).
Who Masked: Outcomes Assessor
Masking Description: Open label, except for the assessors of the primary outcome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bipolar Depression EIPT: Switch to one of the following combinations: (Experimental): Bipolar Depression randomized to EIPT: Switch to 1. one of the following: escitalopram, sertraline, bupropion or venlafaxine plus 2. two of the following: lithium, valproate acid or quetiapine
  Interventions: Drug: Escitalopram; Drug: Sertraline; Drug: Venlafaxine; Drug: Lithium; Drug: Valproate acid; Drug: Quetiapine; Drug: Bupropion
- Bipolar Depression TAU: Switch to quetiapine plus lithium or valproate acid (Active Comparator): Bipolar Depression randomized to TAU: Switch to quetiapine plus lithium or valproate acid Compound, brand, dosage, frequency and duration up to the investigator's discretion (in accordance with SmPC).
  Interventions: Drug: Lithium; Drug: Valproate acid; Drug: Quetiapine

INTERVENTIONS:
Drug: Escitalopram — See arm description
  Other Names: ATC code: N06AB10
  Arms: Bipolar Depression EIPT: Switch to one of the following combinations:
Drug: Sertraline — See arm description
  Other Names: ATC code: N06AB06
  Arms: Bipolar Depression EIPT: Switch to one of the following combinations:
Drug: Venlafaxine — See arm description
  Other Names: ATC code: N06AX16
  Arms: Bipolar Depression EIPT: Switch to one of the following combinations:
Drug: Lithium — See arm description
  Other Names: ATC code: N05AN01
Drug: Valproate acid — See arm description
  Other Names: ATC code: N03AG01
Drug: Quetiapine — See arm description
  Other Names: ATC code: N05AH04
Drug: Bupropion — See arm description
  Other Names: ATC cose: N06AX12
  Arms: Bipolar Depression EIPT: Switch to one of the following combinations:

SUMMARY:
Bipolar disorders affect approximately 4.5 million people across the European Union (EU) and are associated with high annual healthcare and societal costs. Bipolar disorder I and II represent disorders that cause extreme fluctuation in a person's mood, energy, and ability to function, in which symptoms of (hypo)mania and depression alternate. The depressive episodes of bipolar disorders are often referred to as bipolar depression (BD). In other words: it is a phase/state of the disorder. For many patients with BD, the depressive polarity is often more pervasive and more debilitating than manic states, with estimates that depressed mood accounts for up to two-thirds of the time spent unwell, even with treatment. The burden of not received an effective treatment for BD is high: more severe psychopathology, higher rates of unemployment, more hospitalisations, lower quality of life, lower cognitive functioning, risk of suicide, comorbidities and poorer social and occupational functioning and thus more carer burden. For BD, the treatment guidelines are very heterogeneous, amongst other reasons because the disease is heterogeneous and treatments should be tailored to the patients. There is no clear treatment algorithm and it cannot yet be predicted which treatment will be effective. Especially the place of adjunctive antidepressants is under debate. Usually, for psychiatric disorders (including bipolar disorder), a patient is considered to be treatment-resistant is two medicinal treatments have been tried (in sufficient duration and dosage) without sufficient success. For BD, there is no consensus on when to consider a patient as treatment-resistant, but the most common definition is after one prior treatment failure. This raises the research question whether adjunctive antidepressants to treat BD should be introduced earlier in the treatment. Additionally, The INTENSIFY trial is part of the larger Horizon 2021 project, with the central goal of paving the way for a shift towards a treatment decision-making process tailored for the individual at risk for treatment resistance. To that end, we aim to establish evidence-based criteria to make decisions of early intense treatment in individuals at risk for treatment resistance across the major psychiatric disorders of schizophrenia, bipolar disorder and major depression.

DETAILED DESCRIPTION:
Rationale Bipolar disorders affect approximately 4.5 million people across the European Union (EU) and are associated with high annual healthcare and societal costs. Bipolar disorder I and II represent disorders that cause extreme fluctuation in a person's mood, energy, and ability to function, in which symptoms of (hypo)mania and depression alternate. The depressive episodes of bipolar disorders are often referred to as bipolar depression (BD). In other words: it is a phase/state of the disorder. For many patients with BD, the depressive polarity is often more pervasive and more debilitating than manic states, with estimates that depressed mood accounts for up to two-thirds of the time spent unwell, even with treatment. The burden of not received an effective treatment for BD is high: more severe psychopathology, higher rates of unemployment, more hospitalisations, lower quality of life, lower cognitive functioning, risk of suicide, comorbidities and poorer social and occupational functioning and thus more carer burden. For BD, the treatment guidelines are very heterogeneous, amongst other reasons because the disease is heterogeneous and treatments should be tailored to the patients. There is no clear treatment algorithm and it cannot yet be predicted which treatment will be effective. Especially the place of adjunctive antidepressants is under debate. Usually, for psychiatric disorders (including bipolar disorder), a patient is considered to be treatment-resistant is two medicinal treatments have been tried (in sufficient duration and dosage) without sufficient success. For BD, there is no consensus on when to consider a patient as treatment-resistant, but the most common definition is after one prior treatment failure. This raises the research question whether adjunctive antidepressants to treat BD should be introduced earlier in the treatment. Additionally, The INTENSIFY trial is part of the larger Horizon 2021 project, with the central goal of paving the way for a shift towards a treatment decision-making process tailored for the individual at risk for treatment resistance. To that end, we aim to establish evidence-based criteria to make decisions of early intense treatment in individuals at risk for treatment resistance across the major psychiatric disorders of schizophrenia, bipolar disorder and major depression.

Objective The primary objective is to compare the treatment response (baseline; visit 2 vs. end of treatment; visit 4), expressed as symptom severity at six weeks and changes in symptom severity from baseline, as measured through the Montgomery-Åsberg Depression Rating Scale (MADRS) under an early-intensified pharmacological treatment to that under treatment as usual, in subjects who had a first-time treatment failure on their first-line treatment.

Main trial endpoints Change in symptom severity total score from baseline (visit 2) to end of treatment (visit 4). This is measured using MADRS.

Secondary trial endpoints

1. To compare changes in severity and improvement in global functioning assessed by the Clinical Global Impression Scale (CGI) between the two treatment arms.
2. To compare changes in the levels of depression and anxiety between treatment arms.
3. To compare changes in quality of life and functioning measures between treatment arms.
4. To compare changes in cognitive performance between treatment arms.
5. To compare the proportion of participants (EIPT vs. TAU) that is in symptomatic remission at visit 4.
6. To compare presence of side effects between treatment arms.
7. To compare use of concomitant medication between treatment arms.
8. To compare premature discontinuation (timing and reason) between treatment arms.
9. To compare changes in suicidal ideation between treatment arms.
10. To compare occurrence of (hypo)manic episode during the study between the treatment arms.

Trial design The clinical study is an international, multicenter controlled, randomised, open label trial (with blinded raters), with a treatment duration of six weeks.

Trial population The aim is to recruit 418 subjects with bipolar disorder type I or II, currently in a depressive episode. Male and female subjects, in- and out-patients, with the age of at least 18 old are eligible for participation. The main exclusion criteria are defined to protect the wellbeing of subjects, e.g. being pregnant or breastfeeding, subjects with previous failure on quetiapine, meeting any contraindications, or participants with a known intolerance to quetiapine.

Interventions

Subjects are randomised to treatment as usual (second-line treatment) or to the early-intensified pharmacological treatment (third-line treatment). Treatment per can be found in the table below:

Table 1. Overview of treatment randomisation per study sample.

Treatment as Usual (TAU) Switch to quetiapine plus lithium or valproate acid Early-Intensified Pharmacological Treatment (EIPT) Switch to

1. one of the following: escitalopram, sertraline, bupropion or venlafaxine plus
2. two of the following: lithium, valproate acid or quetiapine

Ethical considerations relating to the clinical trial including the expected benefit to the individual subject or group of subjects represented by the trial subjects as well as the nature and extent of burden and risks All medications studied in the current trial are widely used (alone or in combination) in clinical practice and the risks for side effects are well established. In the current study, clinical practice is mimicked as much as possible to maximize generalisability and for feasibility purposes. To this end, Summaries of Product Characteristics (SmPCs) are followed with regards to contraindications (implemented as exclusion criterion), safety measures and allowed combinations with other medications. Site visits and assessments are kept to a minimum to keep subject burden at an acceptable level, while meeting the objectives of the study. Blood samples for biomarker analyses are only collected when subjects provide consent; safety measures are performed as part of clinical routine.

Overall, the risks are similar to daily clinical practice; the only difference relative to clinical practice is the application of three pharmacological treatments (EIPT) versus two (TAU) earlier in the illness. Still, these additional treatment options are also commonly prescribed by clinicians. There are no indications in existing literature or clinical practice that the earlier introduction of these medications poses a safety risk when used in an earlier illness phase than indicated in the SmPC.

A benefit of the study is that if it indeed turns out that the early-intensified treatment is associated with more symptom improvement compared to treatment as usual, future patients have to go through less trial and error, which results in a reduced burden (higher quality of life, less unemployment, less hospitalisations) for patients and carers as well as lower societal and healthcare costs.

IMPORTANT: the study was submitted to the European authorities before (see NCT05603104) and they requested to split this study into 3 studies (1 for each diagnostic category). We have done this and created 3 new ClinicalTrials.gov studies as well, from which this is one for bipolar depression. The ClinicalTrials.gov numbers of the related trials are NCT05958875 for the INTENSIFY SZ trial and NCT05973851 for the INTENSIFY MDD trial. The site in the UK (London) followed the advice and will submit 3 separate protocols and are therefore included in the current record. However, Israel already submitted this as one protocol. Therefore, we keep the old clinicaltrials.gov number for Israel (NCT05603104).

ELIGIBILITY:
Inclusion criteria:

1. In- or out patients, at least 18 years of age.
2. Being willing and able to provide written informed consent. Having a legal guardian to cosign is allowed. Informed consent will be signed at visit 1, before any study procedure.
3. Female subjects of child bearing potential must use effective contraception during the trial as per the requirements of the applicable SmPCs and should have a negative pregnancy test at visit 1 or 2 (before randomisation). Male subjects that will use valproate acid during the trial must use effective contraceptive measures during the trial (see section 8.2.1).
4. Meeting diagnostic criteria for a primary diagnosis of bipolar depression (bipolar disorder type I and II currently in a depressive episode), according to DSM-5. The primary diagnosis will be confirmed by the Mini International Neuropsychiatric Interview (MINI v7.0.2).
5. Subject experiences a treatment failure due to lack of efficacy in the current episode, as confirmed by a CGI-I ≥3; preferably, this treatment is a first-line pharmacotherapeutic agent for the primary DSM-5 diagnosis, and was prescribed for at least 4 weeks within an effective dose range as specified in the Summary of Product Characteristics (SmPCs). However, other lines of treatment are accepted as well.
6. Subject and clinician intend to change pharmacotherapeutic treatment.
7. A minimum symptom severity threshold needs to be present (moderate leve) and subject needs to experience functional impairment.

   * The minimum symptom severity threshold is a score of ≥20 on the Montgomery Åsberg Depression Rating Scale (MADRS)
   * Functional impairment is defined as a score of 5 or higher on any of the three scales of the Sheehan Disability Scale (SDS).

Exclusion criteria

1. Being pregnant or breastfeeding.
2. Subject has a known intolerance to quetiapine or to all EIPT medication or to all TAU medication.
3. Meeting any of the contraindications for quetiapine, or to all EIPT medication or to all TAU medication options, as specified within the applicable SmPC, supported by clinically significant abnormal values on local laboratory tests, electrocardiogram (ECG) or physical examinations.
4. Subject has participated in another clinical trial in which the subject received an experimental or investigational drug or agent within 30 days before visit 1.
5. Subject experiences any other significant disease or disorder which, in the opinion of the investigator, may either put the subjects at risk because of participation in the trial, or may influence the result of the trial, or the subject's ability to participate in the trial.
6. Subjects with active suicidal ideation with some intent to act, without specific plan ("Yes" to question 4 of the Columbia-Suicide Severity Rating Scale (C-SSRS)) or active suicidal ideation with specific plan and intent ("Yes" to question 5 of the C-SSRS), followed by an assessment by the treating clinician who determines it is not safe for the subject to participate in the study.
7. Subject meets criteria for current substance use disorder, as confirmed by the Mini International Neuropsychiatric Interview (MINI v7.0.2). Nicotine dependency is allowed, as well as mild and moderate alcohol and/or cannabis use disorder (as defined by MINI v7.0.2). Severe alcohol and/or cannabis use disorder are not allowed.
8. Subjects have not been committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
9. A score of 12 or higher on the Young Mania Rating Scale (YMRS) in order to exclude subjects with predominant manic symptoms or mixed symptoms.
10. Subjects dependent on the sponsor, investigator or trial site must be excluded from participation in advance.
11. Subjects with pre-existing severe liver damage (as tested within the local laboratory test at visit 1).
12. Subjects with a history of antidepressant-induced mania or hypomania or recent rapid cycling (based on the medical file of the potential participant or the clinical judgment of the clinician).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparing the change in symptom severity on Montgomery Asberg Depression Rating Scale | 6 weeks
  Mean in symptom severity (EIPT vs. TAU) total score from baseline (visit 2) to end of treatment (visit 4). This is measured using the Montgomery Asberg Depression Rating Scale.Minimum score is 0, maximum score is 60. A bigger mean change means a better outcome

SECONDARY OUTCOMES:
Compare proportion of participants that is in symptomatic remission | 6 weeks
  Comparison of the proportion of participants (EIPT vs. TAU) that is in symptomatic remission at visit 4. Remission is defined as a Montgomery Asberg Depression Rating scale score of ≤ 12.
Compare the change in the severity and improvement CGI-S sub-scores | 6 weeks
  To compare changes in the severity sub-score of the Clinical Global Impression Scale (CGI 2) between the two treatment arms (EIPT/TAU) over the six week treatment period (visit 2 versus visit 4). Higher scores indicate higher illness severity. Minimum score: 1, maximum score: 7
Compare the change in the severity and improvement CGI-I sub-scores | 6 weeks
  To compare mean changes in the total improvement sub-score of the Clinical Global Impression (CGI 2) between the two treatment arms (EIPT/TAU) over the six week treatment period (visit 2 versus visit 4). A higher score means lower treatment improvement. Minimum score: 1, maximum score: 7
Compare the changes in the levels of depression and anxiety | 6 weeks
  To compare changes in the levels of depression and anxiety as assessed with the Hospital Anxiety and Depression Scale between the two treatment arms (EIPT/TAU) over the four week treatment period (visit 2 versus visit 4). Lower scores mean less depression and anxiety.
To compare changes in cognitive performance as measured through the Trail Making Test | 6 weeks
  To compare changes in cognitive performance as measured through the Trail Making Test between the two treatment arms over the four weeks treatment period (visit 2 versus visit 4). A lower time to complete the test means better cognitive performance.
To compare the changes in cognitive performance as measured through the Rey Auditory Verbal Learning Test | 6 weeks
  To compare changes in cognitive performance as measured through the Rey Auditory Verbal Learning Test between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4). A higher scores means better cognitive performance.
To compare the changes in subjective cognitive performance as measured through the Perceived Deficits Questionnaire | 6 weeks
  To compare changes in cognitive performance as measured through the Perceived Deficits Questionnaire between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4). A higher scores means worse subjective cognitive performance.
To compare the changes in functioning on the Leuven Affective and Pleasure Scale | 6 weeks
  To compare changes in the functioning measure, Leuven Affective and Pleasure Scale, between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4). A higher scores means worse functioning. Minimum score: 0, Maximum score: 160
To compare the changes in functioning on the Sheehan Disability Scale | 6 weeks
  To compare changes in the functioning measure,Sheehan Disability Scale, between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4). A higher scores means worse functioning. Minimum score: 0, maximum score 30.
To compare the changes in quality of life measure, Quality of Life Enjoyment and Satisfaction Questionnaire Short Form | 6 weeks
  To compare changes in quality of life measure, Quality of Life Enjoyment and Satisfaction Questionnaire Short Form between the two treatment arms over the four weeks treatment period (visit 2 versus visit 4). A higher scores means better quality of life. Minimum score: 16, maximum score: 80.
To compare the changes in quality of life measure, Quality of Life Scale -100, subscale inner tension | 6 weeks
  To compare changes in quality of life measure, Quality of Life Scale -100, subscale inner tension between the two treatment arms over the four weeks treatment period (visit 2 versus visit 4). This is a dichotomous scale (unsatisfactory or satisfactory). More 'satisfactory' answers means higher quality of life.
To compare the frequency of occurence of side effects between the two treatment arms. | 6 weeks
  To compare presence of side effects as measured through General Assessment of Side Effects Scale and reported spontaneously between the two treatment arms (EIPT/TAU) over the six week treatment period (visit 2 versus visit 4). Higher scores means more side effects. Minimum score: 0 side effects, maximum score: 38 side effects.
To compare the proportion of participants using concomitant medication between the two treatment arms. | 6 weeks
  To compare use of concomitant medication between the two treatment arms (EIPT/TAU) over the six week treatment period (visit 2 versus visit 4) effects.
To compare the proportion of participants who prematurely discontinue between the two treatment arms. | 6 weeks
  To compare premature discontinuation between the two treatment arms (EIPT/TAU) over the six week treatment period (visit 2 versus visit 4).
To compare the reason of participants that prematurely discontinue the study treatment between the two treatment arms. | 6 weeks
  To compare the difference in reasons for premature treatment discontinuation between the two treatment arms (EIPT/TAU) over the six week treatment period (visit 2 versus visit 4).
To compare changes in suicidal ideation between treatment arms. | 6 weeks.
  Changes on the Columbia-Suicide Severity Rating Scale (C-SSRS) throughout the study; EIPT vs TAU. Higher score means higher suicidal ideation. Max score is 5.
To compare occurrence of (hypo)manic episode during the study between the treatment arms | 6 weeks.
  Occurrence of (hypo)manic episodes throughout the study (including V5); EIPT vs TAU. Scores of 12 or higher means that a participant is in a (hypo)manic episode of bipolar disorder.

CONTACTS AND LOCATIONS:
Locations (13):
- Medical University Innsbruck, Innsbruck, Austria
- Germany (5):
  - Universitätsklinik für Psychiatrie und Psychotherapie Bielefeld, Bielefeld
  - LWL-Klinik Dortmund, Bereich Forschung & Wissenschaft, Dortmund
  - University Hospital Frankfurt am Main - Goethe University, Frankfurt am Main
  - Klinik für Psychiatrie und Psychotherapie der Universitätsmedizin Mainz, Mainz
  - Westfälische Wilhelms-Universität Münster, Münster
- Eginition hospital, department of psychiatry, Athens, Greece
- Italy (4):
  - Universita degli Studi di Brescia, Brescia
  - University of Cagliari, Cagliari
  - Università degli studi della Campania Luigi Vanvitelli, Naples
  - Azienda Ospedaliero-Universitaria "Città della Salute e della Scienza di Torino", Turin
- Fundació Clínic per a la Recerca Biomèdica, Barcelona, Spain
- King's College London, Psychiatry & Cognitive Neuroscience, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR